CLINICAL TRIAL: NCT03662360
Title: Elderly Patients With Dementia in the Department of Acute Geriatrics: Pilot Study, Monocentric, Randomized Use of Aromatherapy as a Complementary Treatment to Psychopharmacotherapy in Psychological Disorders and BPSD Behavior
Brief Title: Elderly Demented Patients: Aromatherapy Complementary to Psychopharmacotherapy Psychological Disorders and BPSD Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Luganese Moncucco (Other)
Responsible Party: Principal Investigator, Pio Eugenio Fontana, Head of Geriatric Division, Clinica Luganese Moncucco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLM_ds_p_02
Record Dates: First submitted 2018-06-07; First posted 2018-09-07 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: BPSD (Behavioral and Psycological Symptoms of Dementia)
Keywords: BPSD (behavioral and psycological symptoms of dementia); aromatherapy; elderly
MeSH Terms: conditions — Behavior | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: The enrolled patients will be randomized following the 4 blocks random schema (AABB, ABAB, BBAA, BABA, ABBA, BAAB).
  A repetition of the first 4 blocks will be perform up to 32 patients:
  AABB, ABAB, BBAA, BABA AABB, ABAB, BBAA, BABA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A - control group (No Intervention): 16 patients who respect the inclusion criteria, treated with psychotropic drugs Pro Re Nata.
- GROUP B - aromatherapy group (Experimental): 16 patients included in the inclusion criteria, treated with psychotropic drugs Pro Re Nata and, in a complementary way, with diffusion aromatherapy
  Interventions: Other: essential oils

INTERVENTIONS:
Other: essential oils — Following a specific schema, the randomization will be perfomed. Patients enrolled in Group B will receive in environmental diffusion two essential oils, to define their possible effectiveness in the control of the psychological and behavioural disorders
  Other Names: lavander essential oil; wild orange essential oil
  Arms: GROUP B - aromatherapy group

SUMMARY:
Behavioral and psycological symptoms of dementia, (BPSD) are one of the major problem for families, doctors and for patients the same. To reduce the side effects of the standard treatments, is important to find an alternative methods of treatment, eg the aromatherapy. There is an incresing in scientific evidence the its use in dementia behavior related.

DETAILED DESCRIPTION:
Behavioral and psycological symptoms of dementia, (BPSD) are one of the major problem for families, doctors and for patients the same.

In absence of the universally recognized guidelines, the standard treatment involves the use of psychotropic drugs (typical / atypical neuroleptics, antidepressants, benzodiazepines) that are often not very effective and involve a series of side effects such as sedation, slowing down -motor with impaired cognitive performance, cardiac electrical changes and extrapyramidal syndrome. In view of this, it is important to find an alternative methods of treatment, which can reduce psychological and behavioral disorders and at the same time the use of psychotropic drugs.

As for aromatherapy, ie the therapeutic use of natural essential oils, there is a decades-long clinical experience, especially in France, which is accompanied by increasing scientific evidence with considerable increase in publications in its use in psychological disorders and dementia behavior related. Based on the scientific publications available, it was therefore decided to use two essential oils (Citrus sinensis, Lavandula angustifolia) in environmental diffusion in the Geriatric Department of the Clinica Luganese Moncucco.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the acute geriatric ward;
* patients with a known diagnosis of dementia associated with BPSD or diagnosis performed during hospitalization.

Exclusion Criteria:

* patients with alcohol-based dementia;
* patients with Mild Cognitive Impairment (MCI) - section 4 -;
* patients with language barrier;
* patients already being treated with aromatherapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Franzetti Pellanda, MD, Study Director — Clinica Luganese Moncucco; Pio Eugenio Fontana, MD, Study Director — Clinica Luganese Moncucco
Locations (1):
- Clinica Luganese Moncucco, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
A UPN will be attributed to each patient. The dataset containing the correspondence between the UPN and the patient's personal and clinical data will be kept at the Clinical Research Unit of the Clinica Luganese Moncucco. All the analyzed data that will be published or available for scientific discussions will be codified.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after the end of data collection
Access Criteria: All the available data will be codified

REFERENCES:
- [Background] Ballard CG, Gauthier S, Cummings JL, Brodaty H, Grossberg GT, Robert P, Lyketsos CG. Management of agitation and aggression associated with Alzheimer disease. Nat Rev Neurol. 2009 May;5(5):245-55. doi: 10.1038/nrneurol.2009.39. PMID 19488082
- [Background] Margallo-Lana M, Swann A, O'Brien J, Fairbairn A, Reichelt K, Potkins D, Mynt P, Ballard C. Prevalence and pharmacological management of behavioural and psychological symptoms amongst dementia sufferers living in care environments. Int J Geriatr Psychiatry. 2001 Jan;16(1):39-44. doi: 10.1002/1099-1166(200101)16:13.0.co;2-f. PMID 11180484
- [Background] Lonergan E, Luxenberg J, Colford J. Haloperidol for agitation in dementia. Cochrane Database Syst Rev. 2002;(2):CD002852. doi: 10.1002/14651858.CD002852. PMID 12076456
- [Background] Ballard C, Corbett A. Agitation and aggression in people with Alzheimer's disease. Curr Opin Psychiatry. 2013 May;26(3):252-9. doi: 10.1097/YCO.0b013e32835f414b. PMID 23528917
- [Background] Ballard C, Howard R. Neuroleptic drugs in dementia: benefits and harm. Nat Rev Neurosci. 2006 Jun;7(6):492-500. doi: 10.1038/nrn1926. PMID 16715057
- [Background] Schneider LS, Dagerman K, Insel PS. Efficacy and adverse effects of atypical antipsychotics for dementia: meta-analysis of randomized, placebo-controlled trials. Am J Geriatr Psychiatry. 2006 Mar;14(3):191-210. doi: 10.1097/01.JGP.0000200589.01396.6d. PMID 16505124
- [Background] Schneider LS, Tariot PN, Dagerman KS, Davis SM, Hsiao JK, Ismail MS, Lebowitz BD, Lyketsos CG, Ryan JM, Stroup TS, Sultzer DL, Weintraub D, Lieberman JA; CATIE-AD Study Group. Effectiveness of atypical antipsychotic drugs in patients with Alzheimer's disease. N Engl J Med. 2006 Oct 12;355(15):1525-38. doi: 10.1056/NEJMoa061240. PMID 17035647
- [Background] Ballard C, Hanney ML, Theodoulou M, Douglas S, McShane R, Kossakowski K, Gill R, Juszczak E, Yu LM, Jacoby R; DART-AD investigators. The dementia antipsychotic withdrawal trial (DART-AD): long-term follow-up of a randomised placebo-controlled trial. Lancet Neurol. 2009 Feb;8(2):151-7. doi: 10.1016/S1474-4422(08)70295-3. Epub 2009 Jan 8. PMID 19138567
- [Background] Ballard CG, O'Brien JT, Reichelt K, Perry EK. Aromatherapy as a safe and effective treatment for the management of agitation in severe dementia: the results of a double-blind, placebo-controlled trial with Melissa. J Clin Psychiatry. 2002 Jul;63(7):553-8. doi: 10.4088/jcp.v63n0703. PMID 12143909
- [Background] Holmes C, Hopkins V, Hensford C, MacLaughlin V, Wilkinson D, Rosenvinge H. Lavender oil as a treatment for agitated behaviour in severe dementia: a placebo controlled study. Int J Geriatr Psychiatry. 2002 Apr;17(4):305-8. doi: 10.1002/gps.593. PMID 11994882
- [Background] O'Connor DW, Eppingstall B, Taffe J, van der Ploeg ES. A randomized, controlled cross-over trial of dermally-applied lavender (Lavandula angustifolia) oil as a treatment of agitated behaviour in dementia. BMC Complement Altern Med. 2013 Nov 13;13:315. doi: 10.1186/1472-6882-13-315. PMID 24219098
- [Background] Jimbo D, Kimura Y, Taniguchi M, Inoue M, Urakami K. Effect of aromatherapy on patients with Alzheimer's disease. Psychogeriatrics. 2009 Dec;9(4):173-9. doi: 10.1111/j.1479-8301.2009.00299.x. PMID 20377818
- [Background] Elisabetsky E, Marschner J, Souza DO. Effects of Linalool on glutamatergic system in the rat cerebral cortex. Neurochem Res. 1995 Apr;20(4):461-5. doi: 10.1007/BF00973103. PMID 7651584
- [Background] Huang L, Abuhamdah S, Howes MJ, Dixon CL, Elliot MS, Ballard C, Holmes C, Burns A, Perry EK, Francis PT, Lees G, Chazot PL. Pharmacological profile of essential oils derived from Lavandula angustifolia and Melissa officinalis with anti-agitation properties: focus on ligand-gated channels. J Pharm Pharmacol. 2008 Nov;60(11):1515-22. doi: 10.1211/jpp/60.11.0013. PMID 18957173
- [Background] Kim JT, Ren CJ, Fielding GA, Pitti A, Kasumi T, Wajda M, Lebovits A, Bekker A. Treatment with lavender aromatherapy in the post-anesthesia care unit reduces opioid requirements of morbidly obese patients undergoing laparoscopic adjustable gastric banding. Obes Surg. 2007 Jul;17(7):920-5. doi: 10.1007/s11695-007-9170-7. PMID 17894152
- [Background] Barocelli E, Calcina F, Chiavarini M, Impicciatore M, Bruni R, Bianchi A, Ballabeni V. Antinociceptive and gastroprotective effects of inhaled and orally administered Lavandula hybrida Reverchon "Grosso" essential oil. Life Sci. 2004 Nov 26;76(2):213-23. doi: 10.1016/j.lfs.2004.08.008. PMID 15519366
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] de Oliveira AM, Radanovic M, de Mello PC, Buchain PC, Vizzotto AD, Celestino DL, Stella F, Piersol CV, Forlenza OV. Nonpharmacological Interventions to Reduce Behavioral and Psychological Symptoms of Dementia: A Systematic Review. Biomed Res Int. 2015;2015:218980. doi: 10.1155/2015/218980. Epub 2015 Nov 29. PMID 26693477
- [Background] Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD006211. doi: 10.1002/14651858.CD006211.pub3. PMID 28898390
- [Background] Kaufer DI, Cummings JL, Christine D, Bray T, Castellon S, Masterman D, MacMillan A, Ketchel P, DeKosky ST. Assessing the impact of neuropsychiatric symptoms in Alzheimer's disease: the Neuropsychiatric Inventory Caregiver Distress Scale. J Am Geriatr Soc. 1998 Feb;46(2):210-5. doi: 10.1111/j.1532-5415.1998.tb02542.x. PMID 9475452
- [Background] Wood S, Cummings JL, Hsu MA, Barclay T, Wheatley MV, Yarema KT, Schnelle JF. The use of the neuropsychiatric inventory in nursing home residents. Characterization and measurement. Am J Geriatr Psychiatry. 2000 Winter;8(1):75-83. doi: 10.1097/00019442-200002000-00010. PMID 10648298
- [Background] Directive 2001/20/EC of the European Parliament and of the Council of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the member states relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use. Med Etika Bioet. 2002 Spring-Summer;9(1-2):12-9. No abstract available. PMID 16276663
- [Background] Dixon JR Jr. The International Conference on Harmonization Good Clinical Practice guideline. Qual Assur. 1998 Apr-Jun;6(2):65-74. doi: 10.1080/105294199277860. PMID 10386329
- [Background] [The Helsinki Declaration of the World Medical Association (WMA). Ethical principles of medical research involving human subjects]. Pol Merkur Lekarski. 2014 May;36(215):298-301. No abstract available. Polish. PMID 24964504
- See also: details about mild cognitive impairment — http://www.uptodate.com/contents/mild-cognitive-impairment-epidemiology-pathology-and-clinical-assessment?search=mild%20cognitive%20impairment&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NPI NH> or = 1 at T1 (NPI-NH score from 0 to 144, patients with a score from 1 to 144 have been enrolled)
Period: Overall Study
Arm/Group | GROUP A - Control Group | GROUP B - Aromatherapy Group
Started | 16 | 16
Completed | 16 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- GROUP A - Control Group: 16 patients who respect the inclusion criteria, treated with psychotropic drugs.
- GROUP B - Aromatherapy Group: 16 patients included in the inclusion criteria, treated with psychotropic drugs and, in a complementary way, with diffusion aromatherapy
  essential oils: Following a specific schema, the randomization will be perfomed. Patients enrolled in Group B will receive in environmental diffusion two essential oils, to define their possible effectiveness in the control of the psychological and behavioural disorders
- Total: Total of all reporting groups
Arm/Group | GROUP A - Control Group | GROUP B - Aromatherapy Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 1 | 9 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 16 | 16 | 32
patients admitted to the geriatric acute ward in may-june 2018 CLM [Number; unit: participants] | 16 | 16 | 32
patients with diagnosis of dementia associated with BPSD or diagnosis made during hospitalization [Number; unit: participants] | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Role of Essential Oil Therapy in Environmental Diffusion as a Complement of Psychotropic Drugs in the Management of Psychological and Behavioral Disorders (BPSD)
Description: The Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) test will characterize the neuropsychiatric and psychopathological symptoms of patients affected by dementia.
  Events as delirium, anxiety, depression, etc. will be recorded by the frequency (from 0, absence, to 4, high frequency) and the seriousness (from 0, absence, to 3, high). The total score of the NPI-NH is given by the frequency x (multiply) seriousness (total score for each event has a range from 0 to 12). The patient final score will be given by the sum of the score of the 12 events. For each patient will be given a total score from 0 to 144.
  NPI NH score has been collected in both control and aromatherapy groups at T1 and T3, in patients who needed and who did not needed Pro Re Nata.
Time Frame: Time 1 (baseline) and Time 3 (day 7)
Population: All participants with NPI-NH evaluated at Time 1 and Time 3
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | GROUP A - Control Group | GROUP B - Aromatherapy Group
Number analyzed (Participants) | 16 | 14
score on a scale
  T1 NPI score in patients do not need Pro Re Nata | 21.81 [6 to 42] | 25.93 [9 to 60]
  T3 NPI score in patients needed Pro Re Nata: number analyzed (Participants) | 8 | 6
  T3 NPI score in patients needed Pro Re Nata | 32.87 [18 to 51] | 16.5 [9 to 33]
  T3 NPI score in patients do not need Pro Re Nata: number analyzed (Participants) | 8 | 8
  T3 NPI score in patients do not need Pro Re Nata | 20.00 [5 to 42] | 7.25 [5 to 10]
Statistical Analysis 1: Comparison: GROUP A - Control Group vs GROUP B - Aromatherapy Group; The Mann-Whitney test has been used to evaluate the statistical significance of the difference between the variations in scores (T3 - T1) regarding the two interest groups of patients (control and treated); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Role of Essential Oil Therapy in Environmental Diffusion in Professional Caregiver Distress Linked to BPSD
Description: NPI-NH assess the psychological distress in physicians, nurses and nursing assistants who managed the patients. It has a score from 0 (no discomfort) to score of 5 (extreme discomfort). The psychological distress is measured for each of the 12 events in the NPI-NH scale, for a total score from 0 to 60.
Time Frame: Time 1 (baseline) and Time 3 (day 7)
Population: To evaluate the physicians, nurses and nursing assistants distress, both control and aromatherapy group were subdivided into two groups: use or not use of PNR. PNR was used at T3, so the difference between T1 and T3 was a comparison to evaluate the evolution of distress.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | GROUP A - Control Group | GROUP B - Aromatherapy Group
Number analyzed (Participants) | 16 | 14
score on a scale
  T1 NPI NH physicians in pts with PRN: number analyzed (Participants) | 8 | 6
  T1 NPI NH physicians in pts with PRN | 4.19 [0 to 18] | 5.64 [0 to 15]
  T1 NPI NH physicians in pts without PRN: number analyzed (Participants) | 8 | 8
  T1 NPI NH physicians in pts without PRN | 1.60 [0 to 9] | 4.13 [0 to 20]
  T1 NPI NH nurses in pts with PRN: number analyzed (Participants) | 8 | 6
  T1 NPI NH nurses in pts with PRN | 9.63 [0 to 25] | 11.64 [0 to 21]
  T1 NPI NH nurses in pts without PRN: number analyzed (Participants) | 8 | 8
  T1 NPI NH nurses in pts without PRN | 6.40 [0 to 14] | 10.13 [0 to 27]
  T1 NPI NH nursing assistants in pts with PRN: number analyzed (Participants) | 8 | 6
  T1 NPI NH nursing assistants in pts with PRN | 11.00 [0 to 27] | 12.21 [0 to 23]
  T1 NPI NH nursing assistants in pts without PRN: number analyzed (Participants) | 8 | 8
  T1 NPI NH nursing assistants in pts without PRN | 7.10 [0 to 15] | 10.88 [0 to 31]
  T3 NPI NH physician in pts with PRN: number analyzed (Participants) | 8 | 6
  T3 NPI NH physician in pts with PRN | 6.00 [0 to 21] | 2.64 [0 to 15]
  T3 NPI NH physician in pts without PRN: number analyzed (Participants) | 8 | 8
  T3 NPI NH physician in pts without PRN | 3.20 [0 to 12] | 0.88 [0 to 6]
  T3 NPI NH nurses in pts with PRN: number analyzed (Participants) | 8 | 6
  T3 NPI NH nurses in pts with PRN | 12.00 [0 to 27] | 5.79 [0 to 19]
  T3 NPI NH nurses in pts without PRN: number analyzed (Participants) | 8 | 8
  T3 NPI NH nurses in pts without PRN | 9.30 [0 to 19] | 4.25 [0 to 10]
  T3 NPI NH nursing assistants in pts with PRN: number analyzed (Participants) | 8 | 6
  T3 NPI NH nursing assistants in pts with PRN | 13.19 [0 to 28] | 5.93 [0 to 19]
  T3 NPI NH nursing assistants in pts without PRN: number analyzed (Participants) | 8 | 8
  T3 NPI NH nursing assistants in pts without PRN | 9.90 [0 to 19] | 4.38 [0 to 10]
Statistical Analysis 1: Comparison: GROUP A - Control Group vs GROUP B - Aromatherapy Group; The Mann-Whitney test has been used to evaluate the statistical significance of the difference between the variations scores in T3 and T1, concerning the distress of the professional caregivers in the two intereste groups of patients; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 days
Description: no adverse events
Groups:
- GROUP B - Aromatherapy Group: 14 patients included in the inclusion criteria, treated with psychotropic drugs Pro Re Nata and, in a complementary way, with diffusion aromatherapy
  essential oils: Following a specific schema, the randomization will be perfomed. Patients enrolled in Group B will receive in environmental diffusion two essential oils, to define their possible effectiveness in the control of the psychological and behavioural disorders
Arm/Group | GROUP A - Control Group | GROUP B - Aromatherapy Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03662360/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03662360/SAP_001.pdf